CLINICAL TRIAL: NCT02912442
Title: Thyroid Autoimmunity and Reproductive Failure - a Study of Autoimmunity in Association With Treatment Outcome in Infertile Danish Women With Infertility or Recurrent Miscarriages.
Brief Title: Thyroid Autoimmunity and Reproductive Failure in Danish Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ulla Feldt-Rasmussen, Professor, DMSc, Rigshospitalet, Denmark
Other Study IDs: THY-FER-IMM
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Thyroid; Infertility; Autoantibodies; Autoimmunity; Pregnancy Loss
Keywords: thyroid; infertility; autoimmunity; pregnancy loss; autoantibodies
MeSH Terms: conditions — Thyroid Diseases; Infertility; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Infertile women study 1
- Infertile women study 2
- Repeated pregnancy loss

SUMMARY:
The present Ph.D.-study investigates the mechanisms behind the association between thyroid autoimmunity and reproductive failure.

ELIGIBILITY:
Inclusion Criteria:

* Women followed in the Fertility Clinic

Exclusion Criteria:

* Pregnancy at time of blood sampling. Immune-suppressive ⁄modulatory treatments. Women referred for oocyt donation, genetic testing, and hepatitis and HIV-positivity

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women referred to the infertility clinic
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Live birth | 2011-2015

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Undecided